CLINICAL TRIAL: NCT00248690
Title: Intracranial Pressure (ICP) Versus Intracranial Compliance (ICC) Guided Management in Subarachnoid Hemorrhage; - a Prospective, Randomized Trial.
Brief Title: ICP Versus Intracranial Compliance Guided Management in SAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Audun Stubhaug / Professor, Rikshospitalet-Radiumhospitalet HF
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2005-SAHD; S-05184
Record Dates: First submitted 2005-10-25; First posted 2005-11-04 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2008-01

CONDITIONS: Subarachnoid Hemorrhage (SAH)
Keywords: Subarachnoid hemorrhage; Intracranial hypertension; Intracranial pressure; Diagnostic techniques and procedures; Compliance; Treatment outcome; Intensive care, surgical
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Hypertension; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

INTERVENTIONS:
Device: ICP mean wave amplitude — Appropriate measures when ICP mean wave amplitude is to high, e.g. CSF drainage

SUMMARY:
The purpose of this study is to determine whether treatment guided also by ICP mean wave amplitude improves outcome compared to international standard care in patients with SAH.

DETAILED DESCRIPTION:
In this study SAH-patients are randomized to treatment based on international standard care (ICP/CPP guided therapy) or intracranial compliance (ICP mean wave amplitude) guided therapy in addition to ICP/CPP guided therapy. Main outcome variables are survival and neurological outcome after 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage, acute
* Intracerebral pressure monitoring device inserted

Exclusion criteria:

* No intracranial pressure monitoring
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-11; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
All cause mortality and neurological outcome | 3 and 12 months

SECONDARY OUTCOMES:
Length of stay (ICU, hospital); complications; effect of treatment modalities on mean ICP, CPP, ICP mean wave amplitude. | Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Bentsen, MD, Study Director — Oslo University Hospital
Locations (1):
- Rikshospitalet University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Eide PK, Sorteberg A, Bentsen G, Marthinsen PB, Stubhaug A, Sorteberg W. Pressure-derived versus pressure wave amplitude-derived indices of cerebrovascular pressure reactivity in relation to early clinical state and 12-month outcome following aneurysmal subarachnoid hemorrhage. J Neurosurg. 2012 May;116(5):961-71. doi: 10.3171/2012.1.JNS111313. Epub 2012 Feb 10. PMID 22324419